CLINICAL TRIAL: NCT06245863
Title: Measurement and Treatment With Laser and Mechanical Systems to Treat Back Pain
Brief Title: Measurement and Treatment of Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of Minas Gerais (Other)
Collaborators: Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other)
Responsible Party: Principal Investigator, Fernanda Rossi Paolillo, Professor, State University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Back Pain
Record Dates: First submitted 2024-01-19; First posted 2024-02-07 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain | interventions — Lasers; Ultrasonography

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Negative pressure and Laser: Combined Therapy (Experimental): Vacuum therapy combined with laser on back pain.
  Interventions: Device: Negative pressure and Laser
- Positive Pressure and Laser: Combined Therapy (Experimental): Rollers combined with laser on back pain.
  Interventions: Device: Positive Pressure and Laser
- Ultrasound and Laser: Combined Therapy (Experimental): Ultrasound combined with laser on back pain.
  Interventions: Device: Ultrasound and Laser
- Laser (Active Comparator): Infrared Laser on back pain.
  Interventions: Device: Laser
- Placebo Laser (Placebo Comparator): The placebo laser treatment.
  Interventions: Device: Placebo Laser

INTERVENTIONS:
Device: Negative pressure and Laser — Synergistic application (single handle) - Laser: Red (660 nm) and infrared (808 nm) lasers, continuous mode, 100 milliwatts (mW) per laser. Vacuum therapy: 60 mm suction cup, pulsed mode (MP9, 50 pulsations per minute) and pressure of -150 at -350 mbar. The treatment was carried out during 20 minutes on the lumbar, thoracic and cervical spine regions. Seven sessions were performed.
  Arms: Negative pressure and Laser: Combined Therapy
Device: Positive Pressure and Laser — Synergistic application (single handle) - Laser: Red (660 nm) and infrared (808 nm) lasers, continuous mode, 100 mW per laser. Positive Pressure: Massage with rollers. The treatment was carried out during 20 minutes on the lumbar, thoracic and cervical spine regions. Seven sessions were performed.
  Arms: Positive Pressure and Laser: Combined Therapy
Device: Ultrasound and Laser — Synergistic application (single handle) - Laser: Red (660 nm) and infrared (808 nm) lasers, continuous mode, 100 mW per laser. Ultrasound: 1 megahertz (MHz), continuous mode and 1 milliwatts per square centimeter (mW/cm2). The treatment was carried out during 20 minutes on the lumbar, thoracic and cervical spine regions. Seven sessions were performed.
  Arms: Ultrasound and Laser: Combined Therapy
Device: Laser — Infrared Laser (808 nm), continuous mode, 100 mW. The treatment was carried out during 20 minutes on the lumbar, thoracic and cervical spine regions. Seven sessions were performed.
  Arms: Laser
Device: Placebo Laser — Laser: off mode. The placebo treatment was carried out during 20 minutes on the lumbar, thoracic and cervical spine regions. Seven sessions were performed.
  Arms: Placebo Laser

SUMMARY:
The aim of this study was to evaluate the clinical aspects and to investigate the therapeutic effects of combined therapy with laser on back pain.

DETAILED DESCRIPTION:
Dysfunctions of the musculoskeletal system are related to physiological, kinesiological and biomechanical factors that result in pain, paresthesia, inflammation, heaviness, fatigue and compression of peripheral nerves. Clinical aspects related to back pain were investigated. For treatment, photobiomodulation can be performed with laser equipment that emits red and infrared light, which promotes analgesic and anti-inflammatory effects. Mechanical stimulus can be combined with laser to improve therapeutical effects. In this context, the laser was combined with ultrasound, negative pressure and positive pressure to treat back pain.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers (female and male)
* Aged between 20 and 60 years
* Who had medical referral for pain complaint in low back

Exclusion Criteria:

* Psychiatric illnesses
* Endocrinopathies
* Heart diseases
* Neurological diseases
* Osteoporosis
* Cancer
* Analgesic, anti-inflammatory or muscle relaxant drugs in the last four weeks

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 1 day and 7 weeks
  Visual analogue scale (VAS): The volunteer was instructed to give a score for pain intensity between 0 (no pain) and 10 (worst imaginable pain).
Algometry - Pressure threshold measurement | 1 day and 7 weeks
  Pain pressure threshold on low back using algometer. Data obtained in Newton. Higher pressure pain threshold is reported for lower pain sensitivity.
Dynamometry - Strenght measurement | 1 day and 7 weeks
  Isometric trunk strength using dynamometer. Data obtained in Newton. greater the value, greater the strength.

SECONDARY OUTCOMES:
Anamnesis | 1 day
  Questionnaire to get the clinical characteristics of patients.
Body mass index (BMI) measurement | 1 day
  Body mass index: BMI = mass (kg) / height2 (m). Classification: BMI less than 18.5 kg/m2 are underweight, BMI between 18.5 and 24.9 kg/m2 is considered normal weight, BMI between 25 and 29.9 kg/m2 is considered overweight, and BMI ≥ 30 kg/m² is considered obese. Obesity is divided into grades; grade I being a BMI between 30 to 34.9 kg/m², grade II being a BMI 35 to 39.9 kg/m² and grade III BMI ≥ 40 kg/m².
Waist-hip ratio (WHR) measurement | 1 day
  Waist-hip ratio: WHR = waist (cm) / hips (cm). The anatomical landmarks to measure the circumference (cm), in the upright position of the body were: 1) waist: measured at the above the iliac crest; 2) hip: measured at the largest protuberance of the buttocks. Classification: Gynoid (WHR between 0.68 and 0.8) and Android (WHR>0.8).
Body composition measurement | 1 day
  Body composition was performed to evaluate the hydration and the body fat percentage using bipolar bioimpedance.
Shoulder mobility measurement | 1 day and 7 weeks
  Bilateral range of motion was assessed, combining internal rotation with shoulder adduction and external rotation with abduction of the other shoulder, placing the hand on the central axis of the body in the thoracic region. Three distance measurements were obtained on both sides between the third fingers of the right and left hands to calculate the average.
Flexibility of the spine | 1 day and 7 weeks
  Fingertip-to-floor test was carried out. In upright standing position with knees joint fully extended, the volunteers were instructed to bend forward and attempt to reach for the floor with their fingertips. The distance between the patient's right long finger and the floor were measured using a measuring tape. Three measurements were taken to calculate the average value.
Goniometry - Angular measurement | 1 day and 7 weeks
  Active goniometry was performed to assess range of motion (ROM) of the spine (angular measure).
Quality of life assessment | 1 day and 7 weeks
  Quality of Life was measured using the World Health Organization Quality of Life-Abbreviated form (WHOQOL-BREF), a 26-item questionnaire in which items are rated on a 5-point scale. It evaluates 4 domains related to physical factors, psychological factors, social relationships, and environmental context. Higher scores indicate a better quality of life.
Well-being assessment | 1 day and 7 weeks
  The Subjective Well-Being Scale (EBES) was answered by patients. It is composed of 62 items related to three factors that evaluate subjective well-being: positive affect; negative affection and satisfaction with life versus life dissatisfaction. The first 47 items measure positive and negative affect using a 5-point scale with ratings from "not at all" to "to a great extent". The last 22 items measure life satisfaction (or dissatisfaction) using a 5-point scale with ratings from "strongly disagree" to "strongly agree".

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda R Paolillo, PhD, Principal Investigator — State University of Minas Gerais
Locations (1):
- Fernanda Rossi Paolillo, Passos, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paolillo FR, Luccas GAA, Parizotto NA, Paolillo AR, de Castro Neto JC, Bagnato VS. The effects of transcranial laser photobiomodulation and neuromuscular electrical stimulation in the treatment of post-stroke dysfunctions. J Biophotonics. 2023 Apr;16(4):e202200260. doi: 10.1002/jbio.202200260. Epub 2023 Jan 2. PMID 36520347
- [Background] Paolillo FR, Lobo da Costa PH, Mendes PVB, Cruz DMCD, Paolillo AR, Bagnato VS. Effects of the infrared laser on classical ballerinas' feet: Analysis of plantar foot and static balance. J Bodyw Mov Ther. 2021 Apr;26:246-252. doi: 10.1016/j.jbmt.2020.09.007. Epub 2020 Sep 28. PMID 33992253
- [Background] Mroczek B, Lubkowska W, Jarno W, Jaraczewska E, Mierzecki A. Occurrence and impact of back pain on the quality of life of healthcare workers. Ann Agric Environ Med. 2020 Mar 17;27(1):36-42. doi: 10.26444/aaem/115180. Epub 2019 Dec 30. PMID 32208577
- [Background] Salemi MM, Gomes VMDSA, Bezerra LMR, Melo TMS, Alencar GG, Montenegro IHPM, Calado APM, Montenegro EJN, Siqueira GR. Effect of Dry Cupping Therapy on Pain and Functional Disability in Persistent Non-Specific Low Back Pain: A Randomized Controlled Clinical Trial. J Acupunct Meridian Stud. 2021 Dec 31;14(6):219-230. doi: 10.51507/j.jams.2021.14.6.219. PMID 35770601
- [Background] Kenareh R, Mirmohammadi SJ, Khatibi A, Shamsi F, Mehrparvar AH. The Comparison of The Efficacy of Photobiomodulation and Ultrasound in the Treatment of Chronic Non-specific Neck Pain: A Randomized Single-Blind Controlled Trial. J Lasers Med Sci. 2021 May 17;12:e20. doi: 10.34172/jlms.2021.20. eCollection 2021. PMID 34733743